CLINICAL TRIAL: NCT04265716
Title: Topical Lactobacillus Reuteri DSM 17938 to Evaluate Safety and Efficacy on Children With Mild or Moderate Atopic Dermatitis
Brief Title: Topical L. Reuteri in Children With Atopic Dermatitis
Acronym: ADreuteri
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovacion y Desarrollo de Estrategias en Salud (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Pedro Gutierrez Castrellon, Head of Research for Mother-Child, Innovacion y Desarrollo de Estrategias en Salud
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CSUB0174
Record Dates: First submitted 2020-02-09; First posted 2020-02-12 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo controlled trial, 2 parallel arms. Children with mild or moderate atopic dermatitis will be randomly selected at the Pediatric Dermatologic Clinic-Hospital General GEA-Mexico if they fulfill selectioncriteria.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blinded study. All study staff, including the Principal Investigator and the persons performing the subject assessments, will be blinded during the study. Sealed individual treatment code envelopes will be kept at the clinic to be able to break the code if any emergency occurs, as judged by the Investigator. Tubes with interventions has the same exterior appearence. Emollient are similar in consistency and odour
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L. reuteri (Active Comparator): Topical administration of ointment with L. reuteri DSM17938, rubbed into skin twice per day
  Interventions: Other: Topical L. reeuteri
- Placebo (Placebo Comparator): Rubbed into skin twice per day
  Interventions: Other: Topical L. reeuteri

INTERVENTIONS:
Other: Topical L. reeuteri — Tubes with ointment containing L. reuteri DSM17938

SUMMARY:
This study evaluates the safety and efficacy of the probiotic L. reuteri vs control product as an adjuvant for improving the skin appearance of children with mild or moderate atopic dermatitis. All children will receive the standard of care. Half of the children will receive topical L. reuteri in emollient, while the other half will receive the standard of care plus control product

DETAILED DESCRIPTION:
AD if a very frequent allergic skin disorders in children. Produce a negative significant impact on quality of life and related costs. Recently the changes of skin microbiota had been related with inadequate evolution of atopic dermatitis.

L. reuteri had been identified with some effect to reduce skin inflammation and help to modulate inflammatory pathways on skin. Investigators expect using topical L. reuteri as adjuvant some improvement on skin appearance due to the mode of action previous referenced additionally to some potential changes on microbiome

ELIGIBILITY:
Inclusion Criteria:

* Children age 1 to 8 years old
* Atopic Dermatitis (AD) according to the criteria of Hanifin and Rajka
* SCORAD Index 15 to 50, inclusive
* Subjects whose parents or legal representative are willing to sign the informed consent
* When the child is 8, he/she must also give consent to participate in the study

Exclusion Criteria:

* Use of phototherapy for atopic dermatitis
* Systemic or topic corticosteroids in tthe 30 days prior to the study
* Immunosuppressive or cytostatic drugs in the 2 months prior to the study
* Use of probiotics in the 2 weeks prior to the study
* Other allergic severe disease (asthma, allergic rhinitis)
* Systemic antibiotics in the four days prior to the study
* Fever (temperature> 37.5 °C axillary or equivalent)
* Pathologies associated with immunodeficiency or cancer processes
* Dermatological diseases that may hinder the evaluation of atopic dermatitis or require the continued use of topical corticosteroids
* Subjects for whom any of the studies products are contraindicated according to their technical specifications
* Subjects who have participated in research studies with any products in the 3 months prior to the trial

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2020-02-13 (Actual); Primary Completion 2020-05-13 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Skin appearance modification | 16 weeks
  To evaluate the use of a topical emolient containing L. reuteri DSM17938, in terms of its effect on appearance and symptomology in children with mild to moderate atopic dermatitis evaluated by SCORAD test

SECONDARY OUTCOMES:
Frequency of adverse events | 16 weeks
  To evaluate the frequency of adverse events after the use of topical L. reuteri DSM17938
Changes on Quality of life | 16 weeks
  To evaluate the changes in quality of life after the use of topical L. reuteri DSM17938, evaluated by Children's Dermatology Life Quality Index Score
Changes on Family Quality of life: Familys Dermatology Life Quality Index Score | 16 weeks
  To evaluate the changes in quality of life after the use of topical L. reuteri DSM17938, evaluated by Familys Dermatology Life Quality Index Score.
Frecuency of rescue medications | 16 weeks
  To evaluate the improvement on AD control after the use of topical L. reuteri DSM17938 by frequency of rescue medications
Changes on Skin microbiota | 12 weeks
  To evaluate the skin microbiome after the use of topical L. reuteri through genomic analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Dr. Manuel Gea Gonzalez, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amalia N, Orchard D, Francis KL, King E. Systematic review and meta-analysis on the use of probiotic supplementation in pregnant mother, breastfeeding mother and infant for the prevention of atopic dermatitis in children. Australas J Dermatol. 2020 May;61(2):e158-e173. doi: 10.1111/ajd.13186. Epub 2019 Nov 12. PMID 31721162
- [Background] Yang W, Tu R, Hu Y, He T, Zhang W, Gu L, Liu H. Probiotics supplement for the prevention of eczema in children: Study protocol for a meta-analysis and systematic review. Medicine (Baltimore). 2019 Aug;98(34):e16957. doi: 10.1097/MD.0000000000016957. PMID 31441896
- [Background] Yan DC, Hung CH, Sy LB, Lue KH, Shih IH, Yang CY, Chen LC, Sun HL, Lee MS, Chambard J, Tanguy J, Hughes-Formella B, Nutten S, Blanchard C. A Randomized, Double-Blind, Placebo-Controlled Trial Assessing the Oral Administration of a Heat-Treated Lactobacillus paracasei Supplement in Infants with Atopic Dermatitis Receiving Topical Corticosteroid Therapy. Skin Pharmacol Physiol. 2019;32(4):201-211. doi: 10.1159/000499436. Epub 2019 May 22. PMID 31117100
- [Background] Li L, Han Z, Niu X, Zhang G, Jia Y, Zhang S, He C. Probiotic Supplementation for Prevention of Atopic Dermatitis in Infants and Children: A Systematic Review and Meta-analysis. Am J Clin Dermatol. 2019 Jun;20(3):367-377. doi: 10.1007/s40257-018-0404-3. PMID 30465329
- [Background] Navarro-Lopez V, Ramirez-Bosca A, Ramon-Vidal D, Ruzafa-Costas B, Genoves-Martinez S, Chenoll-Cuadros E, Carrion-Gutierrez M, Horga de la Parte J, Prieto-Merino D, Codoner-Cortes FM. Effect of Oral Administration of a Mixture of Probiotic Strains on SCORAD Index and Use of Topical Steroids in Young Patients With Moderate Atopic Dermatitis: A Randomized Clinical Trial. JAMA Dermatol. 2018 Jan 1;154(1):37-43. doi: 10.1001/jamadermatol.2017.3647. PMID 29117309
- [Background] Prakoeswa CRS, Herwanto N, Prameswari R, Astari L, Sawitri S, Hidayati AN, Indramaya DM, Kusumowidagdo ER, Surono IS. Lactobacillus plantarum IS-10506 supplementation reduced SCORAD in children with atopic dermatitis. Benef Microbes. 2017 Oct 13;8(5):833-840. doi: 10.3920/BM2017.0011. Epub 2017 Oct 12. PMID 29022387
- [Background] Wu YJ, Wu WF, Hung CW, Ku MS, Liao PF, Sun HL, Lu KH, Sheu JN, Lue KH. Evaluation of efficacy and safety of Lactobacillus rhamnosus in children aged 4-48 months with atopic dermatitis: An 8-week, double-blind, randomized, placebo-controlled study. J Microbiol Immunol Infect. 2017 Oct;50(5):684-692. doi: 10.1016/j.jmii.2015.10.003. Epub 2015 Nov 27. PMID 26733351